CLINICAL TRIAL: NCT03506191
Title: Pneumonia Due to Stenotrophomonas Maltophilia in Intensive Care Units: a Multicentre Retrospective Study
Brief Title: Pneumonia Due to Stenotrophomonas Maltophilia in ICUs
Acronym: RETROSTENO
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Groupe Hospitalier Pitie-Salpetriere (Other)
Responsible Party: Principal Investigator, Adrien Bouglé, Study director, Groupe Hospitalier Pitie-Salpetriere
Other Study IDs: RETROSTENO
Record Dates: First submitted 2018-04-13; First posted 2018-04-24 (Actual); Last update posted 2018-08-01 (Actual); Status verified 2018-07

CONDITIONS: Pneumonia, Ventilator-Associated; Stenotrophomonas Infection; Critical Illness; Pneumonia, Bacterial
Keywords: Stenotrophomonas maltophilia; Pneumonia; Intensive Care Unit
MeSH Terms: conditions — Pneumonia, Ventilator-Associated; Critical Illness; Pneumonia, Bacterial; Pneumonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Pneumonia is a major cause of ICU admission, or may complicate ICU course. Among the causative pathogens, Stenotrophomonas Maltophilia is a rare pathogen, but affects usually patients with chronic pulmonary co-morbidities, or with long duration of mechanical ventilation and multiples treatment with broad spectrum antimicrobial therapy. However, there are only a paucity of data regarding epidemiology, impact and outcome of Pneumonia due to Stenotrophomonas Maltophilia in critically ill patients.

Primary objective was to study factors associated with mortality in case of Pneumonia due to Stenotrophomonas Maltophilia. Secondary objectives were to describe factors associated with morbidity of Pneumonia due to Stenotrophomonas Maltophilia (duration of mechanical ventilation, ICU length of stay), and to report the characteristics of critically ill patients presenting Pneumonia due to Stenotrophomonas Maltophilia.

ELIGIBILITY:
Inclusion Criteria:

Patients older than 18 years

Documented Stenotrophomonas maltophilia pneumonia:

* Clinical suspicion (≥ two criteria including: fever> 38.5°C, leukocytosis > 10^9/L or leukopenia < 4.10^8/L, purulent tracheobronchial secretions and a new or persistent infiltrate on chest radiography).
* Documented Stenotrophomonas maltophilia positive quantitative culture of a respiratory sample: bronchoalveolar lavage fluid (significant threshold, >10^4cfu/ml) or plugged telescopic catheter (significant threshold, >10^3cfu/ml) or quantitative endotracheal aspirate (significant threshold, >10^6cfu/ml).

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized in Intensive Care Unit and presenting pneumonia due to Stenotrophomonas maltophilia
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-07-30 (Actual); Study Completion 2018-09-30 (Estimated)

PRIMARY OUTCOMES:
Treatment failure | Day 30
  Treatment failure is defined as composite of death and recurrence of pneumonia due to Stenotrophomonas Maltophilia within 30 days of the first episode

SECONDARY OUTCOMES:
Duration of mechanical ventilation | Day 30
  Number of days under mechanical ventilation
Recurrence of pneumonia due to Stenotrophomonas Maltophilia | Day 30
  New onset of pneumonia due to Stenotrophomonas Maltophilia
Mortality | Day 30

CONTACTS AND LOCATIONS:
Overall Officials: Adrien Bouglé, MD, Study Director — APHP; Philippe Guerci, MD, Principal Investigator — CHRU NANCY
Locations (4):
- France (4):
  - Réanimation Polyvalente CHR Metz-Thionville, Metz
  - Department of Anesthesiology and Critical Care Medicine, University Hospital of NANCY, Nancy
  - Department of Anesthesiology and Critical Care Medicine, University Hospital of Strasbourg, Strasbourg
  - Anesthesiology and Critical Care Medicine, Groupe Hospitalier Pitié-Salpêtrière, Paris, Île-de-France Region

REFERENCES:
- [Derived] Guerci P, Bellut H, Mokhtari M, Gaudefroy J, Mongardon N, Charpentier C, Louis G, Tashk P, Dubost C, Ledochowski S, Kimmoun A, Godet T, Pottecher J, Lalot JM, Novy E, Hajage D, Bougle A; AZUREA research network. Outcomes of Stenotrophomonas maltophilia hospital-acquired pneumonia in intensive care unit: a nationwide retrospective study. Crit Care. 2019 Nov 21;23(1):371. doi: 10.1186/s13054-019-2649-5. PMID 31752976